CLINICAL TRIAL: NCT00573586
Title: Investigational Study For the Treatment of Localized (T1c/T2a) Prostate Cancer With High Intensity Focused Ultrasound (HIFU) Using the Sonablate® 500 (SB-500) System in Canada
Brief Title: Treatment of Localized Prostate Cancer With High Intensity Focused Ultrasound Using the Sonablate® 500 System in Canada
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SonaCare Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: USHIFU-CABC-PC002
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU (Other): Completely destroy prostate cancer tissue, without causing damage to the intervening tissue, with a drop in PSA levels to <0.5ng/ml.
  * Result in negative biopsies for evidence of viable malignant cells after the treatment (12 months if Nadir is not reached or PSA rises from Nadir)
  * Safely treat localized prostate cancer patients, with minimal and acceptable adverse effects
  Interventions: Device: Sonablate 500 (SB-500)

INTERVENTIONS:
Device: Sonablate 500 (SB-500) — Sonablate 500 (SB-500)

SUMMARY:
This is an investigational study on the use of high intensity focused ultrasound (HIFU) in the management of localized prostate cancer (T1c/T2a) as a primary non-comparative study.

High intensity focused ultrasound (HIFU) is a non-invasive acoustic ablation technique that uses intersecting, precision focused ultrasound waves to raise the temperature of the target to) 80-90 degrees C in 2-3 seconds, destroying the targeted tissues (prostate cancer). The tissue targeting is highly precise, minimizing collateral damage.

The overall hypothesis is that HIFU with Sonablate can safely, effectively and selectively ablate prostate cancer tissue, resulting in complete tissue necrosis, in patients diagnosed with localized T1c/T2a prostate cancer, with minimal morbidity.

The specific hypothesis is that the Sonablate has the ability to:

* Completely destroy prostate cancer tissue, without causing damage to the intervening tissue, with a drop in PSA levels to <0.5ng/ml.
* Result in negative biopsies for evidence of viable malignant cells after the treatment (12 months if Nadir is not reached or PSA rises from Nadir)
* Safely treat localized prostate cancer patients, with minimal and acceptable adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Male patients with an initial presentation of organ confined prostate cancer;(clinical stages T1c and T2a only)
* Age 40 yrs. and older up to and including age 80 yrs.
* Anesthesia Surgical Assignment (ASA) categories I, II or III only
* PSA levels equal tyo or less than 10ng/ml
* Pre-HIFU Gleason score equal to or less than 7
* Clearly imageable prostate on TRUS
* Prostate total volume less than 40cc with an AP height less than or equal to 4.2cm. (If volume is greater than 40cc or height greater than 4.2 cm, one 3 monthly shot of an LHRH analogue may be provided, followed by re-imaging of the prostate to document total volume below 40cc.)

Exclusion Criteria:

* Large calcification in the area to be treated (>5mm)
* Bleeding disorder as determined by abnormal prothrombin time (INR) and partial thromboplastin time (PTT)
* Pt. on Coumadin or any other anticoagulent, unless their anticoagulation an be temporarily reversed or stopped
* Urinary tract infection unless treated satisfactorily by antibiotics and documented by a sterile urine culture
* Interest in future fertility
* History of allergy to latex
* Inability to visualize the prostate tissue adequately on transrectal ultrasound imaging
* History of treatment for prostate cancer (except for one LHRH analogue "shrinkage shot")
* History of TURP, thermotherapy or urethral stent
* History of any major rectal surgery
* History of inflammatory bowel disease
* History of urinary bladder neck contracture
* History of any other malignancy other than skin cancer. Patients that have had a previous malignancy and no recurrence of that malignancy within the past 5 years will be allowed; (superficial bladder cancer is OK of clear for 2 years)
* Inability to be placed in lithotomy position Prior long term hormonal therapy for prostate cancer (including bilateral orchiectomy).

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
PSA level | PSA level at 30 and 90 days post treatment

CONTACTS AND LOCATIONS:
Overall Officials: George Vrabec, MD, Principal Investigator — Abbotsford Regional Hospital Cancer Center
Locations (1):
- Abbotsford Regional Hospital Cancer Center, Abbotsford, British Columbia, Canada